CLINICAL TRIAL: NCT01744860
Title: Evaluation of Concordance Between the Methods Used in INCa Platforms and the Cobas® 4800 BRAF V600 Mutation Test for Detection of BRAF V600 Mutations in Melanoma in Real Life Setting
Brief Title: Comparison of In-House Methods and Cobas BRAF V600 Mutation Assay in Melanoma Tumor Samples
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28471
Record Dates: First submitted 2012-12-06; First posted 2012-12-07 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2015-11

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- INCa molecular genetics laboratory "in-house" methods: BRAF V600 mutations were analysed using INCa (Institut National du Cancer [French National Cancer Institute]) molecular genetics laboratories using "in-house" methods
- Cobas 4800 Mutation Test: BRAF V600 mutations were analysed using Cobas 4800 mutation test

SUMMARY:
This non-interventional study will compare the Cobas BRAF V600 mutation assay with in-house methods used in molecular laboratories for the assessment of the BRAF mutation status in melanoma tumor samples. No patients will be enrolled in this study. Data will be collected for approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

No patients are enrolled. Use of tumor samples only.

* Histologically proven melanoma tumor sample
* Any type of tumor sample: biopsy or surgical specimen of primary tumor or metastasis
* Tumor samples must be fixed and paraffin-embedded.

Exclusion Criteria:

No patients are enrolled. Use of tumor samples only.

* Fixative unknown

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: No patients are enrolled in this study. Use of melanoma tumor samples.
Sampling Method: Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- France (12):
  - Boulogne-Billancourt
  - Colmar
  - Lille
  - Lyon
  - Marseille
  - Montpellier
  - Nantes
  - Paris
  - Pessac
  - Rouen
  - Vandœuvre-lès-Nancy
  - Villejuif

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 12 December 2012 to 03 April 2013 which evaluated 420 samples for detection of BRAF V600 mutation in France laboratories.
Pre-assignment Details: A total 420 melanoma tumor samples were analysed in 12 platform laboratories in France. The paraffin-embedded tumour samples were taken from biopsy or surgical specimen from the internal or external pathology laboratory.
Groups:
- Melanoma Tumor Sample With BRAF V600 Mutation: BRAF V600 mutations were analysed in melanoma tumor samples using INCa (Institut National du Cancer [French National Cancer Institute]) molecular genetics laboratories using "in-house" methods and Cobas 4800 mutation test
Period: Overall Study
Arm/Group | Melanoma Tumor Sample With BRAF V600 Mutation
Started | 420
Completed | 420
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Biological samples were analysed rather than samples
Arm/Group | Melanoma Tumor Sample With BRAF V600 Mutation
Number analyzed (Participants) | 420
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — This study has analysed sample data rather than participants
  Between 18 and 65 years | NA — This study has analysed sample data rather than participants
  >=65 years | NA — This study has analysed sample data rather than participants
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Total not calculated because data are not available (NA) in one or more arms
  Male | NA — Total not calculated because data are not available (NA) in one or more arms

OUTCOME MEASURES:

1. Primary Outcome: BRAF Mutation Status According to Cobas 4800 BRAF V600 Mutation Test vs. INCa Laboratories Molecular Genetics Laboratories
Description: BRAF V600 mutation status was determined by INCa molecular laboratories "in-house" methods and Cobas 4800 BRAF V600 mutation test. Samples were analysed as V600 mutation, No V600 mutation and Non evaluable. Additionally, the type of V600 mutation (E, K, R, D, E2, other V600 mutation, not specified) was also evaluated only by INCa molecular laboratory "in-house" method.
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis. n = number of samples with BRAF V600 mutation by "in-house method".
Measure: Number; unit: number of samples
Units Other Than Participants: Tumor Samples
Groups:
- INCa Molecular Genetics Laboratory "in House" Methods: BRAF V600 mutations were analysed using INCa (Institut National du Cancer [French National Cancer Institute]) molecular genetics laboratories using "in-house" methods
Arm/Group | INCa Molecular Genetics Laboratory "in House" Methods | Cobas 4800 Mutation Test
Number analyzed (Participants) | 420 | 420
Number analyzed (Tumor Samples) | 420 | 420
number of samples
  BRAF V600 mutation- Yes | 150 | 143
  BRAF V600 mutation - No | 264 | 266
  Non evaluable | 6 | 11
  Type of mutation, V600D, n = 150 | 1 | NA — Type of BRAF V600 mutation could not be detected by this method
  Type of mutation, V600E, n = 150 | 133 | NA — Type of BRAF V600 mutation could not be detected by this method
  Type of mutation, V600K, n = 150 | 14 | NA — Type of BRAF V600 mutation could not be detected by this method
  Type of mutation, V600R, n = 150 | 2 | NA — Type of BRAF V600 mutation could not be detected by this method
Statistical Analysis 1: Comparison: INCa Molecular Genetics Laboratory "in House" Methods vs Cobas 4800 Mutation Test; Kappa coefficient was used to compare the concordance between INCa Molecular Genetics Laboratory "in-house" methods and Cobas 4800 Mutation Test; Test type: Superiority or Other; Kappa coefficient = 0.8611, 95% CI 2-sided [0.8125 to 0.9097]

2. Secondary Outcome: Tumor Sample Characteristics-Type of Tumor Sample
Description: The type of tumor sample used for evaluation of BRAF V600 mutation whether it was a biopsy or surgical specimen were reported
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis
Measure: Number; unit: number of samples
Units Other Than Participants: Tumor Samples
Groups:
- Overall Tumour Samples: A total of 420 melanoma samples (surgical specimens or biopsies of primary tumours or metastases) were included in analysis. The samples were collected either from External pathology laboratories or Internal pathology laboratories
Arm/Group | Overall Tumour Samples
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
number of samples
  Biopsy | 87
  Surgical specimen | 333

3. Secondary Outcome: Tumor Sample Characteristics - Source of Tumor Sample
Description: The source of tumor sample for BRAF V600 mutation detection whether taken from internal or external pathology laboratory were reported
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Number; unit: number of samples
Units Other Than Participants: Tumor Samples
Arm/Group | Overall Tumour Samples
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
number of samples
  External pathology laboratory | 182
  Internal pathology laboratory | 238

4. Secondary Outcome: Type of Pathology Laboratory Performing the Fixation or Embedding-Pre-analytical Method
Description: The external or internal pathology laboratories involved in the process of fixation or embedding of the tumor sample was evaluated.
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Number; unit: number of samples
Units Other Than Participants: Tumor Samples
Arm/Group | INCa Molecular Genetics Laboratory "In-house" Methods
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
number of samples
  External pathology laboratory | 183
  Internal pathology laboratory | 237

5. Secondary Outcome: Time From Sampling to Fixation- Pre-analytical Method
Description: Time taken from the sampling to the fixation of the tumor sample was reported in range of 0-2 hours, 2-6 hours, >6 hours and unknown. Number of samples falling in each of the class were reported.
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Number; unit: number of samples
Units Other Than Participants: Tumor Samples
Arm/Group | INCa Molecular Genetics Laboratory "In-house" Methods
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
number of samples
  0-2 hours | 140
  2-6 hours | 72
  >6 hours | 3
  Unknown | 205

6. Secondary Outcome: Type of Fixative Used- Pre-analytical Method
Description: The different types of fixative Excell, formol, alcohol formol acetic acid and other, used to fix the tumor samples were reported.
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Number; unit: number of samples
Units Other Than Participants: Tumor Samples
Arm/Group | INCa Molecular Genetics Laboratory "In-house" Methods
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
number of samples
  Alcohol Formol Acetic acid (AFA) | 19
  Excell | 10
  Formol | 389
  Other | 2

7. Secondary Outcome: Fixation Duration by Pre-analytical Method
Description: Fixation duration is defined as the amount of time required in hours for the fixation of a samples. The fixation duration was categorized as <6 hours, 6-24 hours and >24 hours and unknown. Number of samples falling in each category were reported
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Number; unit: number of samples
Units Other Than Participants: Tumor Samples
Arm/Group | INCa Molecular Genetics Laboratory "In-house" Methods
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
number of samples
  <6 hours | 25
  6-24 hours | 107
  >24 hours | 82
  Unknown | 206

8. Secondary Outcome: Slice Thickness by Pre-analytical Method
Description: Slice thickness of all the tumour samples was measured. The slice thickness was measured in micrometer.
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Mean (Standard Deviation); unit: micrometer (µm)
Units Other Than Participants: Tumor Samples
Arm/Group | INCa Molecular Genetics Laboratory "In-house" Methods
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
micrometer (µm) | 7.1 (4.2)

9. Secondary Outcome: Dewaxing by Pre-analytical Method
Description: Dewaxing is a method to recover the DNA from samples. Dewaxing information was collected as "Yes, No or Missing"
Time Frame: Up to 6 Months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Number; unit: number of samples
Units Other Than Participants: Tumor Samples
Arm/Group | INCa Molecular Genetics Laboratory "In-house" Methods
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
number of samples
  Missing | 0
  No | 39
  Yes | 381

10. Secondary Outcome: Necrosis Percentage Determination by Pre-analytical Method
Description: The percentage of necrosis defined as the death of one or more cells in the analysed zone was reported.
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis. Only 341 samples out of 420 were analysed as the information on presence of necrosis was missing for 79 samples in the assessed zones.
Measure: Mean (Standard Deviation); unit: percentage
Units Other Than Participants: Tumor Samples
Arm/Group | INCa Molecular Genetics Laboratory "In-house" Methods
Number analyzed (Participants) | 341
Number analyzed (Tumor Samples) | 341
percentage | 3.6 (8.8)

11. Secondary Outcome: Percentage of Tumor Cells by Pre-analytical Method
Description: The percentage of tumor cells in the given tumor sample were reported.
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Mean (Standard Deviation); unit: percentage
Units Other Than Participants: Tumor Samples
Arm/Group | INCa Molecular Genetics Laboratory "In-house" Methods
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
percentage | 70.8 (20.0)

12. Secondary Outcome: Tumor Samples With Presence of Melanin by Pre-analytical Method
Description: The tumor samples with presence of melanin were categorized as Important, Few, Medium and Absent.
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis. Only available samples were included for analysis.
Measure: Number; unit: number of samples
Units Other Than Participants: Tumor Samples
Arm/Group | INCa Molecular Genetics Laboratory "In-house" Methods
Number analyzed (Participants) | 391
Number analyzed (Tumor Samples) | 391
number of samples
  Few | 127
  Medium | 43
  Important | 19
  Absent | 202

13. Secondary Outcome: DNA Extraction - Extraction Method by Pre-analytical Method
Description: This method assessed DNA from the tumor samples was extracted by Automated method or Manual method.
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Number; unit: number of samples
Units Other Than Participants: Tumor Samples
Arm/Group | INCa Molecular Genetics Laboratory "In-house" Methods
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
number of samples
  Automated extraction method | 188
  Manual extraction method | 232

14. Secondary Outcome: Median DNA Elution Volume by Pre-analytical Method
Description: Median DNA elution volume microliters [mcl] was reported.
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Median (Full Range); unit: mcl
Units Other Than Participants: Tumor Samples
Arm/Group | INCa Molecular Genetics Laboratory "In-house" Methods
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
mcl | 100 [25 to 185]

15. Secondary Outcome: Mean DNA Concentration by Pre-analytical Method
Description: The DNA concentration in the tissue elute was measured in nanogram per microliter (ng/mcL).
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Mean (Standard Deviation); unit: ng/mcl
Units Other Than Participants: Tumor Samples
Arm/Group | INCa Molecular Genetics Laboratory "In-house" Methods
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
ng/mcl | 155.25 (206.85)

16. Secondary Outcome: Amount of DNA by Pre-analytical Method
Description: The total DNA concentration extracted from the tissue was measured in nanogram (ng).
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Mean (Standard Deviation); unit: ng
Units Other Than Participants: Tumor Samples
Arm/Group | INCa Molecular Genetics Laboratory "in House" Methods
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
ng | 11816 (14407)

17. Secondary Outcome: Size of Amplicons Used by "In-house" Analytical Method
Description: The method described the size of amplicon used. It was measured in base pairs (bp).
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Median (Full Range); unit: bp
Units Other Than Participants: Tumor Samples
Arm/Group | INCa Molecular Genetics Laboratory "In-house" Methods
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
bp | 120 [70 to 232]

18. Secondary Outcome: Method of Mutation Detection by "In-house" Analytical Method
Description: Allele-specific PCR, High Resolution Melting (HRM) + Sanger sequencing, Pyrosequencing, Sanger sequencing, Real time PCR, SNaPshot were used for BRAF V600 mutation detection.
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Number; unit: number of samples
Units Other Than Participants: Tumor Samples
Arm/Group | INCa Molecular Genetics Laboratory "In-house" Methods
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
number of samples
  Allele-specific PCR | 128
  HRM + Sanger sequencing | 118
  Pyrosequencing | 67
  Real time PCR | 26
  SNaPshot | 30
  Sanger sequencing | 51

19. Secondary Outcome: Number of Samples Punched in In-house Analytical Method
Description: Total number of samples for whom punch was used in 'in-house analytical' method are reported.
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Number; unit: number of samples
Units Other Than Participants: Tumor Samples
Arm/Group | INCa Molecular Genetics Laboratory "In-house" Methods
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
number of samples
  Yes | 117
  No | 303

20. Secondary Outcome: Mean Number of Slices Per Sample Used for "In-house"- Analytical Method
Description: The mean of number of slices per sample when no punch was used are reported.
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis. Data for the samples where the punch was not used were considered for analysis.
Measure: Mean (Standard Deviation); unit: number of samples
Units Other Than Participants: Tumor Samples
Arm/Group | INCa Molecular Genetics Laboratory "In-house" Methods
Number analyzed (Participants) | 303
Number analyzed (Tumor Samples) | 303
number of samples | 2.6 (1.6)

21. Secondary Outcome: Median Time Between Receipt of Samples and Determination of Result by "In-house" Analytical Method
Description: This In-house analytical method measured the time between receipt of samples to the result determination. It measured the time in days.
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Median (Full Range); unit: days
Units Other Than Participants: Tumor Samples
Arm/Group | INCa Molecular Genetics Laboratory "In-house" Methods
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
days | 7 [1 to 30]

22. Secondary Outcome: Technician Work Time Between DNA Extraction and Result by "In-house" Analytical Method
Description: The working time required by the technician from the time of DNA extraction to the time to obtain the results was measured in hours.
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Median (Full Range); unit: hours
Units Other Than Participants: Tumor Samples
Arm/Group | INCa Molecular Genetics Laboratory "In-house" Methods
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
hours | 7 [2 to 28]

23. Secondary Outcome: Mean DNA Concentration as Measured by COBAS 4800 BRAF V600 Mutation Test-Analytical Method
Description: The DNA concentration as assessed by COBAS 4800 BRAF V600 Mutation assay was reported. The unit used to measure the DNA concentration was nanogram/microlitre (ng/mcl)
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Mean (Standard Deviation); unit: ng/mcl
Units Other Than Participants: Tumor Samples
Arm/Group | Cobas 4800 Mutation Test
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
ng/mcl | 64.62 (78.01)

24. Secondary Outcome: Punch Used for Cobas 4800 BRAF V600 Mutation Test- Analytical Method
Description: The punch done during Cobas 4800 BRAF V600 Mutation Test on the sample was described as Yes or No.
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Number; unit: number of samples
Units Other Than Participants: Tumor Samples
Arm/Group | Cobas 4800 Mutation Test
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
number of samples
  Yes | 45
  No | 375

25. Secondary Outcome: Number of Slices Used When No Punch Was Used for Cobas 4800 BRAF V600 Mutation Test- Analytical Method
Description: This describes the Cobas 4800 BRAF V600 Mutation Test, for the mean of number of slices when No punch method, was used. Of the 420 samples, punch was Yes, for 45 samples and punch was No, for 375 samples.
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis. Data for the samples where the punch was No=375, was used for analysis.
Measure: Mean (Standard Deviation); unit: number of samples
Units Other Than Participants: Tumor Samples
Arm/Group | Cobas 4800 Mutation Test
Number analyzed (Participants) | 375
Number analyzed (Tumor Samples) | 375
number of samples | 2.3 (1.6)

26. Secondary Outcome: Median Time Between Receipt of Sample and Determination of Result by Cobas 4800 BRAF V600 Mutation Test -Analytical Method
Description: This analytical method for cobas 4800 BRAF V600 Mutation Test measured the time between receipt of samples to the result determination. It measured the time in days.
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Median (Full Range); unit: days
Units Other Than Participants: Tumor Samples
Arm/Group | Cobas 4800 Mutation Test
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
days | 6 [1 to 98]

27. Secondary Outcome: Technician Work Time Between DNA Extraction and Result by Cobas 4800 BRAF V600 Mutation Test - Analytical Method
Description: This cobas 4800 BRAF V600 Mutation Test analytical method measures the working time required by the technician from the time of DNA extraction to the time to obtain the results. The time duration was measured in hours.
Time Frame: Up to 6 months
Population: All samples meeting the inclusion criteria and not meeting the exclusion criteria were considered for analysis.
Measure: Median (Full Range); unit: hours
Units Other Than Participants: Tumor Samples
Arm/Group | Cobas 4800 Mutation Test
Number analyzed (Participants) | 420
Number analyzed (Tumor Samples) | 420
hours | 5 [1 to 15]

28. Secondary Outcome: Management of Discordance- Method Used to Manage Discordance
Description: Crossing DNA, DNA from In-House method analysed with cobas, SNaPshot, DNA from cobas analysed with In-House method, external site control test, Sanger sequencing, Kit CE-IVD Therascreen RGQ Qiagen, Kit Therascreen RGQ BRAF + Pyrosequencing by another platform (PF), Pyrosequencing, Mutation detection On Another Block, (primitive tumor [prm. tmr]), Sequencing And Therascreen kit (Qiagen) were used for management of discordance between "in-house" method and Cobas 4800 mutation test.
Time Frame: Up to 6 months
Population: The discordant sample population is defined as the samples whose result for BRAF V600 mutation by the "in-house" method did not show similar outcome with the cobas 4800 mutation test.
Measure: Number; unit: number of samples
Units Other Than Participants: Tumor Samples
Groups:
- Discordant Group: This included 28 samples out of 420 samples, whose BRAF V600 mutation results, by INCa "in House" Methods and cobas 4800 BRAF V600 mutation test did not show similar outcome.
Arm/Group | Discordant Group
Number analyzed (Participants) | 28
Number analyzed (Tumor Samples) | 28
number of samples
  Crossing DNA | 7
  DNA from In-House method analysed with cobas | 6
  SNaPshot | 4
  DNA from cobas analysed with In-House method | 2
  External site control test | 2
  Sanger sequencing | 2
  Kit CE-IVD Therascreen RGQ Qiagen | 1
  KIT THERASCREEN RGQ BRAF+PYROSEQ. by other PF | 1
  Pyrosequencing | 1
  Mutation detection on other Block, (prm. tmr) | 1
  Sequencing and Therascreen kit (Qiagen) | 1

29. Secondary Outcome: Management of Discordance-Final Result for BRAF V600 Mutation Detection
Description: The final results obtained by discordance management of the 28 discordant samples were BRAF V600 mutation, No BRAF V600 mutation and Non-evaluable. These results were further assessed by the Investigator and interpreted as final result.
Time Frame: Up to 6 months
Population: as for outcome 28
Measure: Number; unit: number of samples
Units Other Than Participants: Tumor Samples
Groups:
- Final Result- Discordant Samples: This included 28 samples out of 420 samples, whose BRAF V600 mutation results, by INCa "in House" Methods and cobas 4800 BRAF V600 mutation test did not show similar outcome.
Arm/Group | Final Result- Discordant Samples
Number analyzed (Participants) | 28
Number analyzed (Tumor Samples) | 28
number of samples
  BRAF V600 mutation | 19
  No BRAF V600 mutation | 7
  Non evaluable | 2

ADVERSE EVENTS:
Description: As the samples were used instead of participants for analysis there were no serious or non-serious adverse events reported.
Groups:
- INCa Molecular Genetics Laboratory "in House" Methods: BRAF V600 mutations were analysed using INCa (Institut National du Cancer [French National Cancer Institute]) molecular genetics laboratories using in-house methods
Arm/Group | INCa Molecular Genetics Laboratory "in House" Methods | Cobas 4800 Mutation Test
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.